CLINICAL TRIAL: NCT01809912
Title: A PHASE 1, OPEN LABEL, DOSE ESCALATION STUDY TO INVESTIGATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF MG1102 IN PATIENTS WITH SOLID TUMORS
Brief Title: Safety Study of MG1102 in Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG1102_001
Record Dates: First submitted 2012-10-30; First posted 2013-03-13 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2014-01

CONDITIONS: Solid Tumors
Keywords: solid tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Greenstatin (Experimental): Cohort 1 : 6 mg/m2 Cohort 2 : 12 mg/m2 Cohort 3 : 24 mg/m2 Cohort 4 : 48 mg/m2 Cohort 5 : 96 mg/m2 Cohort 6 : 192 mg/m2 28 Day Course Subjects will receive MG1102 (Recombinant human apolipoprotein(a) Kringle V ) by IV administration on Day 0. If no DLTs are observed during the 6 days following the initial infusion, the same dose will be administered once daily for 5 consecutive days followed by a 2-day rest period three times (over 21 days), completing the course on Day 27.
  Additional 21 Day Courses In the absence of a DLT, and in the case of stable disease or better, a subject may continue to receive MG1102 (Recombinant human apolipoprotein(a) Kringle V
  ) on a compassionate use basis at the same dose and regimen .
  Interventions: Drug: Recombinant human apolipoprotein(a) Kringle V

INTERVENTIONS:
Drug: Recombinant human apolipoprotein(a) Kringle V
  Other Names: Greenstatin

SUMMARY:
To investigate the safety and tolerability of a 28 day course of intravenous (IV) MG1102 in patients with solid tumors for which no standard therapy is available.

DETAILED DESCRIPTION:
This is an open-label, Dose Escalation Study, multicenter phase I study to evaluate the safety and tolerability, determine the pharmacokinetics, and obtain preliminary information regarding pharmacodynamics and efficacy of MG1102 in subjects with solid tumor.

Each subject will receive on dose of MG1102 followed by a 6-day rest period. If the initial dose is tolerated, subject will continue with the 21 days of MG1102 administration (5 days on treatment, 2 days off treatment for 3 weeks.) Subjects that have a tumor response as stable disease, may continue therapy on a compassionate use.

Study Duration : for a minimum of 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Solid tumors refractory to conventional therapy or the subject does not tolerate the conventional therapy
* Evaluable disease or at least one measurable tumor mass by a radiographic technique
* Life expectancy ≥3 months
* Suitable for intravenous administration of study medication
* Signed written informed consent
* Adequate bone marrow, renal, and liver function
* Coagulation profile with aPTT and INR, each ≤ 1.5 x ULN
* No evidence of active Hepatitis B or Hepatitis C infection
* Proteinuria <100 mg
* ECOG performance status ≤2
* Female subjects must agree to use contraceptive measures
* Negative serum ß-hCG
* Ability and willingness to comply with the study protocol

Exclusion Criteria:

* Pregnant or lactating women
* Therapy with systemic anticoagulant or antithrombotic agentswithin 7 days prior to first dose
* Hemoptysis within 3 months prior to first dose
* Cytotoxic chemotherapy, immunotherapy, or radiotherapy within 4 weeks prior to first dose
* Surgery or visceral biopsy within 28 days prior to first dose
* Minor surgical procedure performed within 7 days prior to first dose
* Prior exposure to MG1102
* Known history of HIV
* With active bacterial infections and/or receiving systemic antibiotics
* Current or past diagnosis of leukemia
* Known CNS metastases or clinical evidence of CNS
* Non-healing wound within past 2 weeks
* Bleeding diathesis or bleeding within 14 days prior to enrollment
* Clinically significant thrombosis
* Non-malignant GI bleeding, gastric stress ulcerations, or peptic ulcer disease
* History of idiopathic or hereditary angioedema
* History of sickle cell or any hemolytic anemia
* Require hemoglobin, WBC, or platelet transfusion support or use of hematopoietic growth factors within 2 weeks prior to entry
* Uncontrolled hypertension
* History of clinically significant renal disease
* History of significant medical illness of cardiac or CNS disease within the past 6 months
* Treatment with an investigational agent within the longest time frame of either 5 half-lives or 30 days of initiating study drug
* Medical or psychiatric illness
* Recreational substance use or psychiatric illness
* Known hypersensitivity to MG1102 or components of the formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability IV MG1102 | A minimum of 9 weeks
  Adverse events, physical examinations, vital signs, ECGs, clinical laboratory evaluations, lipid profiles

SECONDARY OUTCOMES:
Each subject's serum drug concentration-time data to determine the pharmacokinetic profile of MG1102 | for 25 days
standard clinical serum tumor markers via serum samples to obtain preliminary information regarding the pharmacodynamics of MG1102 | A minimum of 10 weeks
Determination of response assessed by RECIST v1.1 and Choi criteria to obtain preliminary information regarding the efficacy of MG1102 | A minimum of 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: hyunchul chung, dr, Principal Investigator — Yonsei Cancer Center
Locations (1):
- Yonsei Cancer Center, Yonsei University Severance Hospital, Seoul, Seoul, South Korea